CLINICAL TRIAL: NCT06336330
Title: Early Treatment of Heart Failure: a Non-interventional Study Program of Patients With Heart Failure and Initiated on Dapagliflozin (EVOLUTION-HF DEallEF)
Brief Title: Real-world Study on Dapagliflozin Usage in Patients With Heart Failure (HF) in Germany
Acronym: EvolutionHF-DE
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1699R00050
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Heart Diseases; Cardiovascular Diseases; Heart Failure
Keywords: Heart Failure with preserved ejection fraction (HFpEF); Heart Failure with mildly reduced ejection fraction (HFmrEF); Heart Failure with Reduced Ejection Fraction (HFrEF); Dapagliflozin; Real-World
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFpEF: Adult patients with preserved ejection fraction (HFpEF; EF≥50%) who receive treatment with dapagliflozin in accordance with the local dapagliflozin product label for symptomatic chronic heart failure.
- HFmrEF: Adult patients with mildly reduced ejection fraction (HFmrEF; EF 41-49%) who receive treatment with dapagliflozin in accordance with the local dapagliflozin product label for symptomatic chronic heart failure.
- HFrEF: Adult patients with reduced ejection fraction (HFrEF; EF ≤40%) who receive treatment with dapagliflozin in accordance with the local dapagliflozin product label for symptomatic chronic heart failure.

SUMMARY:
Heart failure (HF) is a global, public health issue that affects more than 63 million people worldwide; this burden is expected to increase substantially as the population ages. Despite advancements in treatment, a HF diagnosis still leads to significant morbidity and mortality; there is also an immense impact on patients' health-related quality of life (HRQoL). Dapagliflozin was recently granted approval for heart failure by the European Commission, regardless of ejection fraction and whether the patient has diabetes. Real-world observational data are necessary to describe dapagliflozin use in real-world settings in order to assess treatment patterns, HF symptoms and their impact on physical limitation, HRQoL and work productivity, as well as health care utilization of patients treated with dapagliflozin in this setting under local treatment standard conditions in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years as of study index date; the study index date is date of initiation of treatment with dapagliflozin
* Patient received/receiving treatment with dapagliflozin in accordance with the local dapagliflozin product label for symptomatic chronic heart failure (HF) and at timepoint of dapagliflozin initiation with:

  * preserved ejection fraction (HFpEF; EF≥50%) OR mildly reduced ejection fraction (HFmrEF; EF 41-49%)
  * OR reduced ejection fraction (HFrEF EF ≤40%)
* Patient is enrolled within 14 to 90 days following initiation of dapagliflozin
* Signed and dated informed consent prior to enrolment in the study

Exclusion Criteria:

* Patient should not be enrolled if he/she is less than 14 days or more than 90 days following initiation of dapagliflozin
* Prior treatment with dapagliflozin or other SGLT2i treatment
* Initiation of dapagliflozin outside of the local HF label
* Diagnosis of Type 1 diabetes prior to enrolment
* Current or planned participation in a clinical trial using an investigational medical product for treating HF
* Patient is involved in the planning and/or conduction of the study
* Hypersensitivity to dapagliflozin or to any of the excipients listed in the SmPC

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received treatment with dapagliflozin for HF since 14-90 day before entering the study will be eligible for enrolment by either primary or secondary care healthcare professionals from outpatient settings. All treatment decisions (i.e., dose and duration of treatment) will be at the discretion of the patient's healthcare provider. Patients may have discontinued from dapagliflozin prior to enrolment onto the study, as long as their dapagliflozin initiation was ≥14 days and ≤90 days prior to enrolment onto the study. Data on other parameters may be obtained at the date of initiation of dapagliflozin by extracting this information retrospectively from medical charts. Patients will only be enrolled after they have given consent to participate in the study. It is at the discretion of the physician whether or not to initiate patients on treatment with dapagliflozin and enrol them in the study.
Sampling Method: Non-Probability Sample
Enrollment: 765 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to discontinuation of dapagliflozin | Baseline to 12 months
  Time from dapagliflozin treatment initiation until the time at which participants stop taking the medication for any reason (from the perspective of the prescriber).
Reasons for discontinuation of dapagliflozin | Baseline to 12 months
  Reasons for discontinuation (from the perspective of the prescriber) of patients initiated on dapagliflozin for HF will be described.
Dose changes of dapagliflozin | Baseline to 12 months
  The number of participants with doses changes for dapagliflozin
Number of patients with dapagliflozin treatment interruptions | Baseline to 12 month
  The number of participants who discontinue treatment with dapagliflozin.
Treatment switches from dapagliflozin to other SGLT2i | Baseline to 12 months
  The number of participants who switch from dapagliflozin to another SGLT2i (Sodium-glucose cotransporter-2 inhibitor) treatment for HF.
Time to other heart failure treatment discontinuation | Baseline to 12 months
  Time from initiation of heart failure medication other than dapagliflozin until the time at which participants discontinued treatment with that medication.
Number of other heart failure treatment initiation | Baseline to 12 months
  The number of participants who initiate new heart failure medication other than dapagliflozin.
Number of other heart failure treatment dosage changes | Baseline to 12 months
  The number of participants with dosage changes for heart failure medication other than dapagliflozin.
Number of other heart failure treatment discontinuation | Baseline to 12 months
  The number of participants who discontinue treatment with heart failure medication other than dapagliflozin.
Number of glucose lowering medication initiation | Baseline to 12 months
  The number of participants who initiate new glucose lowering medication other than dapagliflozin.
Number of glucose lowering medication dosage changes | Baseline to 12 months
  The number of participants with dosage changes for glucose lowering medication other than dapagliflozin.
Number of glucose lowering medication discontinuation | Baseline to 12 months
  The number of participants who discontinue treatment with glucose lowering medication other than dapagliflozin.

SECONDARY OUTCOMES:
Absolute change from baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Measured at 3, 6, 9 and 12 months
  The KCCQ is a 23-item questionnaire that quantifies physical limitations, self-efficacy, social interference and quality of life. Several summary scores may be calculated including: Total Symptom score (measuring symptom frequency and symptom burden), Physical limitation score (measuring limitations in common physical activities), Clinical Summary score (measure of physical limitations and total symptoms), and an Overall Summary score (measure of physical limitations, total symptoms, HRQoL, and social limitations). Summary scores will be examined at each assessment point during follow-up.
Absolute change from baseline in Medication Adherence Report Scale (MARS)-5 questionnaire | Measured at 3, 6, 9 and 12 months
  The MARS-5 is five-item self-report adherence scale which assesses both intentional and non-intentional non-adherence. Respondents rate the frequency with which the five different medication-taking behaviours occur, scoring each item on a 1-5-point scale with higher scores indicating higher reported adherence. The MARS-5 has been shown to be reliable and valid across a variety of health conditions, including cardiovascular and pulmonary diseases.
Absolute change from baseline in Work Productivity and Activity Impairment (WPAI) score | Measured at 3, 6, 9 and 12 months
  The WPAI is a validated instrument to measure impairments in paid and unpaid work and activities. It measures absenteeism (work time missed), presenteeism (impairment at work / reduced on-the-job effectiveness) as well as the impairments in unpaid activity because of health problems during the past seven days. It has been validated to quantify work impairments for numerous diseases such as asthma, psoriasis, irritable bowel syndrome, and Crohn's disease, but has not yet been validated for use in heart failure participants. Scores will be derived from the overall work impairment at each timepoint and then changes of from baseline will be reported.

OTHER OUTCOMES:
The absolute change from baseline in occurrence of depressions in patients initiated on dapagliflozin for HF as captured by the Patient Health Questionnaire-9 (PHQ-9) | Measured at 3, 6, 9 and 12 months
  The PHQ-9 comprises 9 items that capture depressed mood and anhedonia. It has been validated as a screening tool with good evidence of responsiveness. The PHQ-9 score is obtained by adding the score for each question (total points). PHQ-9 score ≥10 showed a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 have been shown to represent mild, moderate, moderately severe, and severe depression, respectively.
Healthcare resource utilisation - Number of hospitalisations since dapagliflozin initiation | Measured at 3, 6, 9 and 12 months
  The number of patients hospitalised will be examined at each assessment point.
Healthcare resource utilisation - Length of HF-related hospital stay since dapagliflozin initiation | Measured at 3, 6, 9 and 12 months
  Duration of outpatient clinic visits in days, will be examined at each assessment point.

CONTACTS AND LOCATIONS:
Locations (43):
- Germany (43):
  - Research Site, Aachen
  - Research Site, Alsfeld
  - Research Site, Bamberg
  - Research Site, Bechhofen
  - Research Site, Bergisch Gladbach
  - Research Site, Berlin
  - Research Site, Brilon
  - Research Site, Bruchsal
  - Research Site, Chemnitz
  - Research Site, Dinslaken
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Frankenthal
  - Research Site, Gera
  - Research Site, Hamburg
  - Research Site, Hoppegarten
  - Research Site, Kaiserslautern
  - Research Site, Kitzingen
  - Research Site, Ludwigsburg
  - Research Site, Ludwigshafen am Rhein
  - Research Site, M Hldorf
  - Research Site, Markkleeberg
  - Research Site, Meiningen
  - Research Site, Münster
  - Research Site, Naumburg
  - Research Site, Nuremberg
  - Research Site, Oschersleben
  - Research Site, Papenburg
  - Research Site, Pirna
  - Research Site, Potsdam
  - Research Site, Querfurt
  - Research Site, Ratingen
  - Research Site, Rostock
  - Research Site, Schleswig
  - Research Site, Schwandorf in Bayern
  - Research Site, Schwäbisch Hall
  - Research Site, Siegen
  - Research Site, Steinfurt
  - Research Site, Stollberg
  - Research Site, Straubing
  - Research Site, Stuttgart
  - Research Site, Ulm
  - Research Site, Wermsdorf

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home